CLINICAL TRIAL: NCT03345225
Title: A Randomized Clinical Study of Precision TACE (P-TACE) With Surefire Infusion Catheter Versus Standard Endhole Catheter (E-TACE) Utilizing Radiopaque Drug Eluting Beads (LUMI) in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: A Clinical Study of Precision TACE (P-TACE) With Surefire
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Miami (Other)
Collaborators: Surefire Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Shree Venkat, M.D., Assistant Professor of Clinical Interventional Radiology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 20170185
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Chemoembolization (TACE); HCC; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Active Comparator): Participants will be randomized to receive DEB-TACE utilizing a standard endhole microcatheter
  Interventions: Device: Standard Endhole Microcatheter
- Surefire Group (Experimental): Participants will be randomized to receive DEB-TACE utilizing the Surefire Infusion System
  Interventions: Device: SureFire Infusion System

INTERVENTIONS:
Device: SureFire Infusion System — Surefire is a modified microcatheter with an expandable cone at its tip to prevent retrograde reflux of flow and change flow dynamics downstream.
  Arms: Surefire Group
Device: Standard Endhole Microcatheter — A Microcatheter with a single hole at the end for a infusion.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to learn about 2 types of FDA-approved catheters used in angiographic (X-ray of blood vessels, with radiopaque substance) procedures like DEB-TACE treatment. The Principal Investigator will check the beads given during the DEB-TACE. They will compare the way in which they are spread out in the tumor and density (how condensed something is).

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years with confirmed diagnosis of unresectable hepatocellular carcinoma who are candidates for TACE therapy
2. Barcelona Clinic Liver Cancer Classification (BCLC) A or B
3. Child-Pugh Class A or B
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. 1 to 5 target tumors that are < 6cm with at least one tumor ≥ 3cm in size
6. Vessel size ≥ 1.5 mm
7. Subject must be able to provide written informed consent

Exclusion Criteria:

1. Extra-hepatic spread of the cancer
2. Macrovascular tumor invasion
3. Diffuse HCC (>50% liver involvement)
4. Previous chemotherapy, radiotherapy, transarterial embolization or ablations in the targeted tumor(s)
5. Advanced liver disease (bilirubin > 3 mg/dl, aspartate aminotransferase (AST) or ALT > 5x upper limit of normal or > 250 U/I
6. Extrahepatic supply to the tumor
7. Hypovascular tumors
8. Heart failure with reduced ejection fraction or Left Ventricular Ejection Fraction (LVEF) ≤ 40 percent
9. Any serious medical or psychiatric illness/condition that will interfere or limit compliance with study requirements/treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Comparing the change in the Lencioni score between the SureFire infusion system and a standard endhole microcatheter | 1 month
  The Lencioni score (calculated by comparing pre and post embolization CT attenuation of the tumor averaged over tumor volume) is used to compare the distribution of chemoembolic beads in the tumor to see if the Surefire Infusion system improves tumor coverage.

SECONDARY OUTCOMES:
The Lencioni Score (LS) | 3 months
  The Lencioni score (calculated by comparing pre and post embolization CT attenuation of the tumor averaged over tumor volume) is used to compare the distribution of chemoembolic beads in the tumor to see if the Surefire Infusion system improves tumor coverage.
The Lencioni Score (LS) | 6 months
  The Lencioni score (calculated by comparing pre and post embolization CT attenuation of the tumor averaged over tumor volume) is used to compare the distribution of chemoembolic beads in the tumor to see if the Surefire Infusion system improves tumor coverage.
Objective Response Rate as measured by mRECIST | 1 Month
  Objective Response Rate (ORR) is the proportion of patients who are responders as confirmed with partial response (PR) or confirmed complete response (CR) based on enhancement pattern and size of target lesions
Objective Response Rate as measured by mRECIST | 3 Month
  Objective Response Rate (ORR) is the proportion of patients who are responders as confirmed with partial response (PR) or confirmed complete response (CR) based on enhancement pattern and size of target lesions
Objective Response Rate as measured by mRECIST | 6 Month
  Objective Response Rate (ORR) is the proportion of patients who are responders as confirmed with partial response (PR) or confirmed complete response (CR) based on enhancement pattern and size of target lesions
Distribution of Radiopaque beads | 1 Month
  Qualitative assessment of the coverage distribution of radiopaque beads, measured on a Likert scale (with response values ranking from 1-5 where 1 is complete coverage and 5 is minimal coverage) in the two treatment arms
Distribution of Radiopaque beads | 3 Month
  Qualitative assessment of the coverage distribution of radiopaque beads, measured on a Likert scale (with response values ranking from 1-5 where 1 is complete coverage and 5 is minimal coverage) in the two treatment arms
Distribution of Radiopaque beads | 6 Month
  Qualitative assessment of the coverage distribution of radiopaque beads, measured on a Likert scale (with response values ranking from 1-5 where 1 is complete coverage and 5 is minimal coverage) in the two treatment arms
Tumor enhancement | 1 month
  Comparing tumor enhancement relative to a calibrated imaging phantom
Tumor enhancement | 3 month
  Comparing tumor enhancement relative to a calibrated imaging phantom
Tumor enhancement | 6 month
  Comparing tumor enhancement relative to a calibrated imaging phantom
Number of Adverse Event | 6 months
  Adverse Event measured by Common Terminology Criteria for Adverse Event (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Shree Venkat, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No